CLINICAL TRIAL: NCT06988254
Title: Animation-Based Breathing Therapy for Children: A Novel Approach for School Settings
Brief Title: Animation-Based Breathing Therapy for School-Age Children
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Tansu Birinci, Principal Investigator, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 17052025
Record Dates: First submitted 2025-05-17; First posted 2025-05-23 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Children; Breathing Patterns; Stress; School Health
Keywords: Children; Breathing; Stress; School; Well-being
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Animation-based breathing therapy (Experimental): The intervention includes the animation-based breathing therapy for six weeks (two sessions per day, five days per week).
  Interventions: Other: Animation-based breathing therapy
- Control (No Intervention): No Intervention

INTERVENTIONS:
Other: Animation-based breathing therapy — The animation-based breathing therapy includes breathing exercises for children, such as lion, crab, and rainbow breathing. The intervention will continue for six weeks (two sessions per day, five days per week).
  Arms: Animation-based breathing therapy

SUMMARY:
This randomized controlled trial aims to investigate the efficacy of animation-based breathing therapy on the physical (cough strength, chest expansion, and walking speed) and psychological health (perceived stress level, well-being, and attention) of school-age children.

DETAILED DESCRIPTION:
One hundred thirty school-age children, aged between 8 and 12, will be randomly assigned to one of two groups: an animation-based breathing therapy group or a control group. The intervention group will receive animation-based breathing therapy for six weeks (two sessions per day, five days per week). Assessments will be conducted at baseline and at the end of the six-week period. Cough strength will be measured using a peak expiratory flow meter. Chest expansion will be assessed with a measuring tape at the axillary, epigastric, and subcostal levels. Walking speed will be evaluated using the 10-Meter Walk Test. Perceived stress will be assessed using the Perceived Stress Scale for Children, well-being will be measured using the WHO-5 Child Wellbeing Index, and attention will be assessed using the Bourdon Attention Test.

ELIGIBILITY:
Inclusion Criteria:

-- Children aged between 8 and 12 years,

* Attending school and formal education regularly,
* Volunteers whose parents and themselves agreed to participate after being informed about the purpose of the study and the procedures involved, and who provided written informed consent.

Exclusion Criteria:

* Children with any condition that may prevent them from completing self-reported questionnaires during the assessment (e.g., difficulty in understanding forms, physical disabilities, illiteracy),
* History of any upper or lower extremity injury within the past six months,
* History of any upper or lower extremity surgery within the past six months,
* Presence of any soft tissue disorder,
* Diagnosed with serious gastrointestinal, cardiovascular, pulmonary, or hematological disorders following examination by a specialist physician,
* Diagnosed spinal problems such as scoliosis, kyphosis, or kyphoscoliosis,
* Diagnosed with psychotic disorder, bipolar disorder, or autism spectrum disorder,
* History of epilepsy or serious head trauma,
* Current use of psychotropic medications.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 130 (Estimated)
Dates: Start 2025-05-20 (Actual); Primary Completion 2025-06-27 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Chest Expansion Measurement | Baseline
  Chest expansion will be assessed using a measuring tape. While the children are in a relaxed seated position, measurements will be taken from the axillary, epigastric, and subcostal regions. The difference between the chest circumference at maximal inspiration and maximal expiration will be calculated and recorded.

SECONDARY OUTCOMES:
Chest Expansion Measurement | After six-week period
  Chest expansion will be assessed using a measuring tape. While the children are in a relaxed seated position, measurements will be taken from the axillary, epigastric, and subcostal regions. The difference between the chest circumference at maximal inspiration and maximal expiration will be calculated and recorded.
Peak Expiratory Flow | Baseline
  Peak expiratory flow will be measured using a peak expiratory flow meter. The children will be instructed to take a deep breath and then exhale as forcefully and as quickly as possible into the device while in a standing position. The highest value from three consecutive trials will be recorded for analysis.
Peak Expiratory Flow | After six-week period
  Peak expiratory flow will be measured using a peak expiratory flow meter. The children will be instructed to take a deep breath and then exhale as forcefully and as quickly as possible into the device while in a standing position. The highest value from three consecutive trials will be recorded for analysis.
10-Meter Walk Test | Baseline
  Walking speed will be assessed using the 10-Meter Walk Test (10MWT). The 10MWT is a performance-based measure used to evaluate walking ability or gait speed over a short distance, expressed in meters per second. A 14-meter walkway will be marked, with 2-meter acceleration and deceleration zones at each end and a central 10-meter section for timing. Children will be asked to walk at their comfortable walking speed. Timing will begin when the child crosses the 2-meter mark and will stop when they pass the 12-meter mark. The time taken to walk the middle 10 meters will be recorded. The average of three trials will be calculated for analysis.
10-Meter Walk Test | After six-week period
  Walking speed will be assessed using the 10-Meter Walk Test (10MWT). The 10MWT is a performance-based measure used to evaluate walking ability or gait speed over a short distance, expressed in meters per second. A 14-meter walkway will be marked, with 2-meter acceleration and deceleration zones at each end and a central 10-meter section for timing. Children will be asked to walk at their comfortable walking speed. Timing will begin when the child crosses the 2-meter mark and will stop when they pass the 12-meter mark. The time taken to walk the middle 10 meters will be recorded. The average of three trials will be calculated for analysis.
Perceived Stress Scale in Children | Baseline
  Perceived stress levels of the children will be assessed using the "Perceived Stress Scale in Children." The scale consists of 9 items, rated on a 4-point Likert scale ranging from 1 (never), 2 (sometimes), 3 (often), to 4 (always). Higher scores indicate higher levels of perceived stress, and there are no reverse-coded items in the scale. The total score ranges from a minimum of 9 to a maximum of 36.
Perceived Stress Scale in Children | After six-week period
  Perceived stress levels of the children will be assessed using the "Perceived Stress Scale in Children." The scale consists of 9 items, rated on a 4-point Likert scale ranging from 1 (never), 2 (sometimes), 3 (often), to 4 (always). Higher scores indicate higher levels of perceived stress, and there are no reverse-coded items in the scale. The total score ranges from a minimum of 9 to a maximum of 36.
WHO-5 Child Wellbeing Index | Baseline
  Children's well-being will be assessed using the WHO-5 Child Wellbeing Index developed by the World Health Organization. The index consists of five positively worded items that reflect the participant's feelings over the past two weeks. Each item is rated on a 6-point Likert scale ranging from 0 to 5, where 0 indicates the absence of positive feelings during the past two weeks, and 5 indicates the constant presence of such feelings. The raw score is calculated by summing the scores of the five items, resulting in a total score between 0 and 25. To obtain a percentage score ranging from 0 to 100, the raw score is multiplied by 4. A score of 0% represents the worst possible well-being, whereas a score of 100% indicates the best possible well-being.
WHO-5 Child Wellbeing Index | After six-week period
  Children's well-being will be assessed using the WHO-5 Child Wellbeing Index developed by the World Health Organization. The index consists of five positively worded items that reflect the participant's feelings over the past two weeks. Each item is rated on a 6-point Likert scale ranging from 0 to 5, where 0 indicates the absence of positive feelings during the past two weeks, and 5 indicates the constant presence of such feelings. The raw score is calculated by summing the scores of the five items, resulting in a total score between 0 and 25. To obtain a percentage score ranging from 0 to 100, the raw score is multiplied by 4. A score of 0% represents the worst possible well-being, whereas a score of 100% indicates the best possible well-being.
Bourdon Attention Test | Baseline
  Attention will be assessed using the Bourdon Attention Test. In this test, children are asked to identify and mark specific target letters within a sequence of randomly arranged letters. A total of 660 letters are presented on a single page, divided into three sections. Participants are given four minutes to complete the task. During this period, they are instructed to locate and mark the designated letters (e.g., a, b, d, g) as quickly and accurately as possible. Scoring is based on the number of correctly marked target letters. Each correct identification is awarded one point, and the total number of accurate responses constitutes the individual's attention score.
Bourdon Attention Test | After six-week period
  Attention will be assessed using the Bourdon Attention Test. In this test, children are asked to identify and mark specific target letters within a sequence of randomly arranged letters. A total of 660 letters are presented on a single page, divided into three sections. Participants are given four minutes to complete the task. During this period, they are instructed to locate and mark the designated letters (e.g., a, b, d, g) as quickly and accurately as possible. Scoring is based on the number of correctly marked target letters. Each correct identification is awarded one point, and the total number of accurate responses constitutes the individual's attention score.

CONTACTS AND LOCATIONS:
Overall Officials: Tansu Birinci Olgun, PT, PhD, Principal Investigator — Istanbul Medeniyet University
Locations (1):
- Istanbul Medeniyet University, Istanbul, Kartal, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided